CLINICAL TRIAL: NCT05013970
Title: Transcatheter Arterial Embolization as a Treatment for Knee Pain in Patients With Mild to Moderate Osteoarthritis
Brief Title: Transcatheter Arterial Embolization in Patients With Mild to Moderate Osteoarthritis
Acronym: Embolization
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial agreement could be found for this study
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S62757
Record Dates: First submitted 2021-08-12; First posted 2021-08-20 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Catheter-directed embolotherapy; Poly-vinyl alcohol microspheres
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Phantoms, Imaging

STUDY DESIGN:
Intervention Model Description: Patients with mild to moderate knee osteoarthritis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee osteoarthritis (Other): Patients with mild to moderate osteoarthritis who suffer from persistent knee pain treated with catheter-directed geniculate artery embolization
  Interventions: Other: Clinical assessment; Other: Radiographic imaging

INTERVENTIONS:
Other: Clinical assessment — Clinical assessment including Visual Analog Scale (VAS) for Knee Pain, and Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire
Other: Radiographic imaging — MRI of the knee

SUMMARY:
Disabling symptoms of osteoarthritis are seen in approximatively 10% of people over 55 years old. Many patients suffer from persistent pain symptoms from moderate osteoarthritis despite optimal medical treatment. For these patients, several minimally-invasive surgical treatments have been proposed, including arthroscopic lavage and debridement; however, none of these treatments have been proven effective compared to sham treatment.

Recently, catheter-directed embolotherapy of the geniculate arteries has been propagated as a real alternative to medical management in patients with mild to moderate knee osteoarthritis unresponsive to conservative medical management.

DETAILED DESCRIPTION:
Disabling symptoms of osteoarthritis are seen in approximatively 10% of people over 55 years old. Traditionally, treatment of symptomatic knee osteoarthritis is based on administration of pain relievers, including nonsteroidal anti-inflammatory drugs, in case of mild to moderate symptoms; major joint replacement surgery (total joint arthroplasty) is performed in cases of severe and end-stage osteoarthritis.

However, many patients suffer from persistent pain symptoms from moderate osteoarthritis despite optimal medical treatment. For these patients, several minimally-invasive surgical treatments have been proposed, including arthroscopic lavage and debridement; however, none of these treatments have been proven effective compared to sham treatment.

Recently, catheter-directed embolotherapy of the geniculate arteries has been propagated as a real alternative to medical management in patients with mild to moderate knee osteoarthritis unresponsive to conservative medical management.

Transcatheter embolotherapy was performed using imipenem/cilastin sodium or 75 micron calibrated Embozene microspheres and follow-up was performed by physical examination, questionnaires (VAS-score and WOMAC-scores) and MR-imaging (WORMS-score). Results of these trials confirmed that catheter-directed embolotherapy is a safe procedure without any major adverse events. WOMAC pain scores dropped dramatically from 12.2 +/- 1.9 before the procedure to 3.3 +/- 2.1 at 1 month after the procedure and to 1.7 +/- 2.2 at 4 months after the procedure. Additionally, MR imaging at 2 years of follow-up could not demonstrate any osteonecrosis or progression of degenerative changes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of knee pain
* Kellgren-Lawrence (KL) grade 1-3 assessed by weight-bearing knee radiographs
* Local tenderness around the knee
* Clinical failure after 3 months or more of conservative therapies, including oral nonsteroidal anti-inflammatory drugs and/or oral opioid agents and physical therapy, stretching, muscle strengthening and/or intra-articular injection of hyaluronic acid
* Persistent moderate to severe knee pain (VAS > 50 mm) for more than 3 months
* Patient is able to give consent

Exclusion Criteria:

* Previous knee surgery
* Local infection
* BMI > 40 kg/m2
* Advanced atherosclerosis
* Rheumatoid arthritis, malignancy, renal insufficiency, other conditions contra-indicating femoropopliteal angiography
* Usage of anticoagulants such as eliquis or coumarine (Asaflow allowed)
* Allergy to iodinated contrast medium or any other allergy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Knee Pain | Within 30 days after catheter-directed embolization
  To measure pain in patients with knee osteoarthritis
Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire | Within 30 days after catheter-directed embolization
  To evaluate symptoms and limitations in patients with knee osteoarthritis
MRI imaging | At day 30 after catheter-directed embolization
  To depict potential asymptomatic, but radiologically visible side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Geert Maleux, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No